CLINICAL TRIAL: NCT05131802
Title: Bile Reflux Gastropathy: Prevalence and Risk Factors After Therapeutic Biliary Interventions: A Retrospective Cohort Study
Brief Title: Bile Reflux Gastropathy: Prevalence and Risk Factors After Therapeutic Biliary Interventions
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Amira Ahmed Othman, Dr., Zagazig University
Other Study IDs: Bile Reflux
Record Dates: First submitted 2021-11-09; First posted 2021-11-23 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Dyspepsia; Heartburn; Bile Reflux
Keywords: Bile Reflux; Cholecystectomy; ERCP; Bilirubin
MeSH Terms: conditions — Dyspepsia; Heartburn; Bile Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Postcholecystectomy group: which included patients that had undergone cholecystectomy.
  Interventions: Device: upper GIT endescopy
- Biliary intervention group: included patients who had undergone at least one of the following procedures for treatment of benign pathology: endoscopic sphincterotomy (ES) and endoscopic stenting.
  Interventions: Device: upper GIT endescopy

INTERVENTIONS:
Device: upper GIT endescopy — Gastric mucosa alterations as erythema, bile existence in the stomach, gastric folds thickening, erosions, and petechiae were also recorded (Olympus single-channel CLK-4). Multiple biopsies were taken from gastric mucosa for histopathological study. Via Triple Lumen ERCP Cannula, 5 mL of gastric fluid was aspirated through the suction channel of the endoscope and collected in a sterile trap placed in the suction line, to be sent for analysis. Quantitative determination of gastric aspirate total bilirubin level was performed (Gen.3® kit and Cobas 8000 analyzer). The pH monitoring of gastric aspirate was performed during the gastroscopy just after collection with a glass electrode pH meter (Adwa®).

SUMMARY:
Bile reflux gastropathy is caused by the backward flow of duodenal fluid into the stomach. A retrospective cohort study was performed to declare if the therapeutic biliary interventions cause bile reflux gastropathy, and to estimate its prevalence and risk factors, and to evaluate the gastric mucosa endoscopic and histopathologic changes.

DETAILED DESCRIPTION:
Bile reflux gastropathy is a pathological condition in the form of the backward flow of duodenal fluid that consists of bile, pancreatic juices, and secretions of the intestinal mucosa into the stomach and esophagus, causing mucosal lesions. Bile acids, in combination with gastric acid, have been shown to cause bile reflux gastropathy symptoms (heartburn, regurgitation, epigastric pain, etc.).

Bile reflux gastropathy frequently occurs after gastric surgeries that that damages the pyloric sphincter, and after biliary surgeries and procedures as cholecystectomy, endoscopic sphincterotomy (EST), endoscopic stenting, or choledochoduodenostomy that cause the sphincter of Oddi malfunction.[4] Bile gastropathy is a normal physiological event in a prolonged fasting period (primary bile reflux gastropathy).In non-responsive individuals to PPI medication, the total prevalence of biliary reflux was 68.7%. These people have acid and bile reflux at the same time and have never had biliary surgery.

Endoscopic retrograde cholangiopancreatography (ERCP) became an increasingly popular modality for both the diagnosis and the treatment of biliary tract disorders. It represents one of the most demanding and technically challenging procedures in gastrointestinal endoscopy, which must be performed effectively and safely by operators with substantial training and experience to maximize success and safety. Cholecystectomy is a surgical operation of gallbladder removal. It can be performed either laparoscopically, using a video camera, or via an open surgical technique. Pain and complications caused by gallstones are the most common reasons for cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Postoperative patients (months to years Postcholecystectomy (Group 1) and therapeutic biliary procedures (Group 2) with persistent upper GIT symptoms ( heartburn, regurgitation dysphagia , dyspepsia ,nausea and epigastric pain) and/or GERD symptoms with history of poor response to prokinetics, mucosa-protective medicines, H2-blockers and/or proton-pump inhibitors (PPI).

Exclusion Criteria:

* included unstable cardiopulmonary, neurologic, or cardiovascular status, other causes of biliary diseases (CBD strictures, and hepatolithiasis), structural abnormalities of the esophagus, stomach, or small intestine, patients who underwent bariatric surgery out of the scope of the study, patients on long-term non-steroidal analgesics, and patients on oral contraceptive drugs.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who were admitted to the university hospitals with inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 288 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
gastric mucosa endoscopic changes as erythema, bile existence in the stomach, gastric folds thickening, erosions, and petechiae. | 7 minutes for endoscopy
  Upper GIT endoscopy is performed and by which gastric mucosa changes were recorded; as erythema, bile existence in the stomach, gastric folds thickening, erosions, and petechiae.
gastric mucosa histopathological changes as chronic inflammation, foveolar hyperplasia , chronic Atrophic gastritis, bile stasis, interstitial inflammation, edema, intestinal metaplasia, and acute inflammation. | 7 minutes for endoscopy for biopsy taken
  Upper GIT endoscopy is performed and by which gastric mucosal biopsies were taken from lesion sites for histopathological study, as chronic inflammation, foveolar hyperplasia , chronic Atrophic gastritis, bile stasis, interstitial inflammation, edema, intestinal metaplasia, and acute inflammation.
intragastric total bilirubin level | 10 minutes for endoscopy for gastric fluid collection
  Upper GIT endoscopy is performed and gastric fluid is aspirated for quantitative analysis of gastric aspirate total bilirubin level
gastric juice pH | 10 minutes for endoscopy for gastric fluid collection
  Upper GIT endoscopy is performed and gastric fluid is aspirated to detect gastric juice pH

CONTACTS AND LOCATIONS:
Overall Officials: Amira A Othman, Ph. D, Principal Investigator — Zagazig University Hospitals
Locations (1):
- Zagazig University Hospitals, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No
to keep participant privacy

REFERENCES:
- [Result] Eldredge TA, Myers JC, Kiroff GK, Shenfine J. Detecting Bile Reflux-the Enigma of Bariatric Surgery. Obes Surg. 2018 Feb;28(2):559-566. doi: 10.1007/s11695-017-3026-6. PMID 29230622
- [Result] Vere CC, Cazacu S, Comanescu V, Mogoanta L, Rogoveanu I, Ciurea T. Endoscopical and histological features in bile reflux gastritis. Rom J Morphol Embryol. 2005;46(4):269-74. PMID 16688361
- [Result] Sun D, Wang X, Gai Z, Song X, Jia X, Tian H. Bile acids but not acidic acids induce Barrett's esophagus. Int J Clin Exp Pathol. 2015 Feb 1;8(2):1384-92. eCollection 2015. PMID 25973022
- [Result] Kuran S, Parlak E, Aydog G, Kacar S, Sasmaz N, Ozden A, Sahin B. Bile reflux index after therapeutic biliary procedures. BMC Gastroenterol. 2008 Feb 11;8:4. doi: 10.1186/1471-230X-8-4. PMID 18267026
- [Result] Monaco L, Brillantino A, Torelli F, Schettino M, Izzo G, Cosenza A, Di Martino N. Prevalence of bile reflux in gastroesophageal reflux disease patients not responsive to proton pump inhibitors. World J Gastroenterol. 2009 Jan 21;15(3):334-8. doi: 10.3748/wjg.15.334. PMID 19140233